CLINICAL TRIAL: NCT03459183
Title: Effects of Non-audible Infra- and Ultrasound on Brain Structure and -Function, Cognitive Functions, and Well-being
Brief Title: Effects of Infra- and Ultrasound on the Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SonicBrain01
Record Dates: First submitted 2018-02-02; First posted 2018-03-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Brain Function; Ultrasound; Cognitive Function; Well-being; Depression; Sleep
MeSH Terms: conditions — Depression | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not know their group assignment (ultrasound - verum, ultrasound - placebo; infrasound - verum, infrasound - placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Infrasound - verum (Experimental): In this condition, participants are exposed with non-audible infrasound from the Infrasound (85dB; 6Hz) source, for 8 constant hours during their night sleep. The source is placed close to the participant's bed (approximately 1-2 meters).
  Interventions: Device: Infrasound (85 dB; 6Hz) source
- Infrasound - placebo (Placebo Comparator): In this condition, participants are not exposed to any sound. The infrasound dummy source is placed close to the participant's bed, exactly like in the Infrasound - verum condition (1-2 meters). The Infrasound dummy source looks exactly like the active infrasound source but produces no sound at all. Participants are told that this source emits sound for 8 constant hours during their night sleep.
  Interventions: Device: Infrasound dummy source
- Ultrasound - verum (Experimental): In this condition, participants are exposed to non-audible ultrasound, emitted by the Ultrasound (10dB below hearing threshold; 22.4 kHz) source for 8 constant hours during their night sleep. The source is placed close to the participant's bed (1-2 meters), at the level of the participant's head (for instance on a nightstand).
  Interventions: Device: Ultrasound (10dB below hearing threshold; 22.4 kHz) source
- Ultrasound - placebo (Placebo Comparator): In this condition, participants are not exposed to any sound. The Ultrasound dummy source is placed close to the participant's bed, exactly like in the Infrasound - verum condition (1-2 meters). The Ultrasound dummy source looks exactly like the active ultrasound source, but produces no sound at all. Participants are told that this source emits sound for 8 constant hours during their night sleep.
  Interventions: Device: Ultrasound dummy source

INTERVENTIONS:
Device: Infrasound (85 dB; 6Hz) source — the infrasound source will emit inaudible 6Hz sound for 8 consecutive hours during participant's night sleep, local sound pressure (at participants head) will be calibrated at 85 dB
  Arms: Infrasound - verum
Device: Ultrasound (10dB below hearing threshold; 22.4 kHz) source — the ultrasound source will emit inaudible 22.4 kHz sound for 8 consecutive hours during night sleep
  Arms: Ultrasound - verum
Device: Infrasound dummy source — the infrasound dummy source looks exactly like the according verum infrasound source but produces absolutely no sound
  Arms: Infrasound - placebo
Device: Ultrasound dummy source — the ultrasound dummy source looks exactly like the according verum ultrasound source but produces absolutely no sound
  Arms: Ultrasound - placebo

SUMMARY:
Findings in neuroscientific research show that the environment one lives in has measurable effects on brain morphology and functioning. Human exposure to airborne infra- and ultrasound has been constantly increasing during the last decades. For instance, the European Renewable Energy Directive, established in 2009, lead to an increased use of wind turbines, generating infrasound. The EU Directive states that until 2020 a 20% of the EUs' total energy needs is to be generated with renewables, therefore the current infrasound load in the European environment will increase further. Similarly, ultrasound is ubiquitous in the modern public environment, emitted from public address systems, animal repellents, industrial machines, even toothbrushes. The present study aims to investigate potential long-term effects of exposure to infra- and ultrasound on subjective well-being, cognitive and brain functioning, as well as on brain structure. The study will apply a randomized-(placebo) controlled single-blind approach to investigate this subject.

DETAILED DESCRIPTION:
Regarding effects of infra- and ultrasound on the brain, a pioneer study demonstrated that exposure to non-audible infrasound was associated with changes of neural activity across several brain regions, including areas involved in auditory and emotional processing, as well as autonomic control. These findings indicate that subliminal infrasound may have pathogenic effects. Research also indicates that low intensity focused ultrasound (LIFU) modulates the BOLD signal. However, the impact of ultrasound on auditory and other brain regions remains broadly unclear until today. Regarding adverse effects of low frequency noise on (mental) health and cognitive functions, preliminary evidence (summarized by two reviews) suggests mainly negative effects on sleep, stress levels (both subjective and objective; i.e. cortisol levels), headaches, fatigue, concentration, and memory. These reviews do however not explicitly address audible low frequency noise vs. non-audible infrasound.

Research on the effects of infra- and ultrasound on cognitive functioning and well-being is in the fledgling stage. The few studies published so far vary strongly in their applied methods and results. Repeatedly, the media has covered stories about individuals suffering from 'ultrasound-sickness', a condition where the affected person suffers from headache, nausea and pain. In line with these subjective accounts, a review paper suggested that ultrasound exposure can be associated with hyperthermia, nausea, headaches, tinnitus and low blood pressure, as well as with neural excitability, irritation, memory problems and difficulties with concentration and learning, suggesting adverse effects of ultrasound exposure regarding (mental) health and cognition.

Nonetheless, there are also indicators of positive effects of these types of sound; a study suggested that brief bursts of infrasound may have a positive effect on cognitive function. Also, pioneer works in the field are currently testing ultrasound therapy for Alzheimer's patients. It appears, that the effects (positive vs. negative) may be highly variable; depending upon the frequency, sound pressure levels and duration of exposure; as well as the quality of sound (mixed audible and non-audible vs. purely non-audible). Future studies need to clearly define these variables in order to be able to make clear statements about effects.

The present study will hopefully shed further light on the long-term effects of (non-audible) infra- and ultrasound regarding human brain connectivity, structure and function, related cognitive functions and overall well-being. This may also lead to a more sophisticated and fact-based debate about 'noise pollution' of modern human living-environments.

Healthy participants, who gave their written consent, will be exposed to infra- or ultrasound for 28 consecutive days during their night sleep. The sound sources produce sound that is at least 10 dB below the hearing threshold. The sources were designed to mimic exposure to infra- and ultrasound in everyday life. The construction and calibration of the sources was realized by experts of the Physical Technical Federal Institute of Germany (Physikalisch Technische Bundesanstalt; PTB), located in Braunschweig. Sound sources will be installed and gauged at the participants' bedrooms, following a standardized procedure and emit sound for 8 hours during the participants' typical sleeping time. N = 60 participants will be randomized to one out of four conditions:

1. Infrasound verum (n = 20; frequency = 6Hz, sound pressure = 85dB)
2. Infrasound placebo (n = 10)
3. Ultrasound verum (n = 20; frequency = 22.4 kHz, sound pressure = variable +/- 10 dB)
4. Ultrasound placebo (n = 10); (single blind procedure).

First, participants, age 18-40, will be screened for eligibility. In addition, a hearing assessment will be conducted to assure normal auditory ability of all participants. Before and after the sound exposure period, participants will be tested using psychological and (neuro-)cognitive test batteries and questionnaires in order to assess psychiatric and somatic symptoms, well-being and cognitive functioning (particularly tasks that also represent everyday cognitive challenges and assess executive functions); (T1, T2). Furthermore, sensitivity to sound (including to infra- and ultrasound) and current exposure to different sound sources (T1 and T2) will be assessed with questionnaires. In addition, Magnet Resonance Imaging (MRI) will be conducted in order to illuminate morphological and functional brain changes (T1 and T2). In the scanner, participants will execute a spatial n-back task. The task assesses participants' working memory and is also suited to assess stressful reactions due to permanent cognitive load - thus constituting a 'proxy' for a stressful working task in real life. During the n-back task, a dot is presented sequentially at different positions in a grid. Participants are instructed to indicate whether the currently presented dot coincides with the dot presented 3 trials before for each of the presented dots. During the 4-week exposure period through infra-/ ultrasound, participants will also fill out weekly questionnaires, assessing well-being, general health levels, psychiatric and somatic symptoms, quality of sleep, headache and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants
* age 18-40
* informed consent for all parts of the study (including MRT)
* none of the exclusion criteria (see below) fulfilled
* normal hearing

Exclusion Criteria:

* age < 18 or > 40 years
* pregnancy or breastfeeding
* living with young children (0-3 years)
* pets in sleeping room (e.g. cats, dogs, rodents, reptiles)
* living at extremely loud/ noisy street
* tinnitus
* chronic disease/ infection of ENT region
* ear deformation/ ear surgery
* (partial) deafness
* hearing aid/ cochlea implant
* degenerative or inflammatory diseases of the central nervous system
* severe cognitive/ neuropsychological impairment
* severe pain syndrome or other severe organic diseases
* epilepsy
* (past or present) psychiatric disorders
* neurological disorders
* severe diabetic polyneuropathy
* malignancies/ cancer
* cardiac insufficiency
* arterial hypertension
* heart attack/ stroke
* severe hepatic or renal insufficiency
* diseases of the hemopoietic system
* alcoholism/ drug addiction
* medical history of severe allergic or toxic reactions
* current participation in drug trial
* doubts about legal capacity/ capability of understanding
* referral to institutions based on court/ official order
* treatment with centrally acting medication (e.g. antipsychotics, antiepileptics, antidepressants, etc.)
* non-removable metal pieces (aneurysm clips, artificial limbs, etc.) or implanted electronic devices (pacemaker, osmotic or other implanted pumps, cochlear implants, etc.)
* claustrophobia
* acute (respiratory) infection, physical uneasiness
* tattoos in the head region, permanent make-up
* non-removable piercings

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Changes in functional connectivity (functional Magnet Resonance Imaging; fMRI) | at baseline (day 0) and after exposure to infra-/ ultrasound (day 28+)
  exploratory analyses of functional brain changes (fMRI) through infra- and ultrasound (verum conditions vs. placebo conditions)
Changes in brain structure (MRI) | at baseline (day 0) and after exposure (day 28+)
  exploratory analyses of structural brain changes (MRI) through infra- and ultrasound (verum conditions vs. placebo conditions)
Changes in depression levels | at baseline (day 0) and after exposure (day 28+)
  changes in Beck's Depression Inventory - II - revised sum scores, indicating a worsening or improvement (increase or decrease in sum scores) of depression through infra- and ultrasound (verum conditions vs. placebo conditions).
Changes in 'vigilance' attentional test score | at baseline (day 0) and after exposure (day 28+)
  worsening or improvement in the maintenance of attention over a prolonged period of time (this is operationalized as a decrease or increase in the number of correct responses; minimum = 0, maximum = 36; assessed by TAP - Test of Attentional Performance: subtest 'vigilance') through infra- and ultrasound (verum conditions vs. placebo conditions).
Changes in memory test score | at baseline (day 0) and after exposure (day 28+)
  worsening or improvement in memory performance (as indicated by the total score in the fMRI spatial n-back task, defined as the absolute number of correct responses [i.e. correct identification of overlapping dot position; minimum of correct responses = 0, maximum = 100], a decrease indicates worsened spatial memory, an increase indicates improved spatial memory; through infra- and ultrasound (verum conditions vs. placebo conditions).
Changes in alertness task score | at baseline (day 0) and after exposure (day 28+)
  worsening or improvement in 'alertness' (as indicated by mean reaction time [RT] to target stimuli; higher mean RT indicates lowered alertness = worsening; lower mean RT indicates improvement in alertness, [TAP - Test of Attentional Performance; subtest 'alertness']), through infra- and ultrasound (verum conditions vs. placebo conditions).
Changes in sleep quality | at baseline (day 0) and after exposure (day 28+)
  worsening or improvement in self-reported sleep quality (decreases or increases in sum score of the Pittsburgh Sleep Quality Index) through infra- and ultrasound (verum conditions vs. placebo conditions).

SECONDARY OUTCOMES:
Changes in somatization (physical health) | at baseline (day 0) and after exposure (day 28+)
  worsening or improvement of self-reported somatization, including cardiovascular, gastrointestinal and respiratory symptoms, as assessed via the sum score of the Brief Symptom Inventory 'somatization' subscale (increases indicate more somatization, decreases indicate less somatization; scale range for the sum score is minimum = 0; maximum = 28) through infra-/ ultrasound (vs. placebo conditions).

CONTACTS AND LOCATIONS:
Overall Officials: Christian Koch, Dr., Study Chair — Physikalisch-Technische Bundesanstalt, Braunschweig, Germany
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Klinik und Poliklinik für Psychiatrie und Psychotherapie, Hamburg, Germany, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weichenberger M, Bauer M, Kuhler R, Hensel J, Forlim CG, Ihlenfeld A, Ittermann B, Gallinat J, Koch C, Kuhn S. Altered cortical and subcortical connectivity due to infrasound administered near the hearing threshold - Evidence from fMRI. PLoS One. 2017 Apr 12;12(4):e0174420. doi: 10.1371/journal.pone.0174420. eCollection 2017. PMID 28403175
- [Background] Weichenberger M, Kuhler R, Bauer M, Hensel J, Bruhl R, Ihlenfeld A, Ittermann B, Gallinat J, Koch C, Sander T, Kuhn S. Brief bursts of infrasound may improve cognitive function--an fMRI study. Hear Res. 2015 Oct;328:87-93. doi: 10.1016/j.heares.2015.08.001. Epub 2015 Aug 7. PMID 26260309
- [Background] Yoo SS, Kim H, Min BK, Franck E, Park S. Transcranial focused ultrasound to the thalamus alters anesthesia time in rats. Neuroreport. 2011 Oct 26;22(15):783-7. doi: 10.1097/WNR.0b013e32834b2957. PMID 21876461
- [Background] Baliatsas C, van Kamp I, van Poll R, Yzermans J. Health effects from low-frequency noise and infrasound in the general population: Is it time to listen? A systematic review of observational studies. Sci Total Environ. 2016 Jul 1;557-558:163-9. doi: 10.1016/j.scitotenv.2016.03.065. Epub 2016 Mar 17. PMID 26994804
- [Background] Leventhall, G., Pelmear, P., and Benton, S., 2003, A review of published research on low frequency noise and its effects: Department for Environment, Food and Rural Affairs.
- [Background] Smagowska B, Pawlaczyk-Luszczynska M. Effects of ultrasonic noise on the human body-a bibliographic review. Int J Occup Saf Ergon. 2013;19(2):195-202. doi: 10.1080/10803548.2013.11076978. PMID 23759188
- [Derived] Ascone L, Kling C, Wieczorek J, Koch C, Kuhn S. A longitudinal, randomized experimental pilot study to investigate the effects of airborne ultrasound on human mental health, cognition, and brain structure. Sci Rep. 2021 Mar 12;11(1):5814. doi: 10.1038/s41598-021-83527-z. PMID 33712644